CLINICAL TRIAL: NCT03568942
Title: A Phase IIa Single-Center, Open-Label Study Evaluating the Pharmacokinetics of Repeat Oral Doses of Gepotidacin (GSK2140944) in Adult Female Participants With Uncomplicated Urinary Tract Infection (Acute Cystitis)
Brief Title: Pharmacokinetic Study of Oral Gepotidacin (GSK2140944) in Subjects With Uncomplicated Urinary Tract Infection (Acute Cystitis)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Biomedical Advanced Research and Development Authority (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 206899
Record Dates: First submitted 2018-06-11; First posted 2018-06-26 (Actual); Results first posted 2020-01-07 (Actual); Last update posted 2020-06-29 (Actual); Status verified 2020-06

CONDITIONS: Infections, Bacterial
Keywords: gepotidacin; GSK2140944; acute cystitis; pharmacokinetics; urinary tract infections
MeSH Terms: conditions — Bacterial Infections; Urinary Tract Infections | interventions — gepotidacin

STUDY DESIGN:
Intervention Model Description: Subjects will receive 1500 mg gepotidacin tablets BID via oral route for 5 days.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Female subjects with acute cystitis (Experimental): Adult female subjects with suspected acute cystitis based on clinical presentation and pyuria (>=10 WBC/mm^3 or presence of leukocyte esterase) and/or nitrite will be included. Subjects will be administered 1500 mg gepotidacin BID for 5 days via the oral route.
  Interventions: Drug: Gepotidacin

INTERVENTIONS:
Drug: Gepotidacin — Gepotidacin tablets will be available at a dose strength of 750 mg. Tablets will be administered BID with water after consumption of food.

SUMMARY:
Gepotidacin (GSK2140944) is a novel triazaacenaphthylene bacterial type II topoisomerase inhibitor that is being developed for the treatment of uncomplicated urinary tract infections (UTIs; acute cystitis). This Phase IIa study will evaluate plasma and urine pharmacokinetics of gepotidacin in female subjects with acute cystitis. Eligible female subjects will receive twice daily (BID) dose of gepotidacin 1500 milligram (mg) for 5 days via oral route. Pre-treatment and post-treatment samples for pharmacokinetic (PK) assessments will be collected throughout the study. The total duration of the study is approximately 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be >=18 to <=65 years of age inclusive, at the time of signing the informed consent.
* The subject has 2 or more of the following clinical signs and symptoms of acute cystitis with onset <=72 hours of the screening assessment: dysuria, frequency, urgency, or lower abdominal pain.
* The subject has pyuria (>=10 white blood cells per cubic millimeters [WBC/mm^3] or the presence of leukocyte esterase) and/or nitrite from a pretreatment clean-catch midstream urine sample based on local laboratory procedures.
* The subject is female. A female subject is eligible to participate if she is not pregnant, not breastfeeding, and at least 1 of the following conditions applies: a) Not a woman of childbearing potential (WOCBP) OR b) A WOCBP who agrees to follow the contraceptive guidance from the Baseline Visit through completion of the Test of Cure (TOC) Visit.
* Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and protocol.

Exclusion Criteria:

* The subject resides in a nursing home or dependent care-type facility.
* The subject has a body mass index >=40.0 kilogram per square meter (kg/m^2) or a body mass index >=35.0 kg/m^2 with obesity-related health conditions such as high blood pressure or uncontrolled diabetes.
* The subject has a history of sensitivity to the study treatment, or components thereof, or a history of a drug or other allergy that, in the opinion of the investigator or medical monitor, contraindicates her participation.
* The subject is immunocompromised or has altered immune defenses that may predispose the subject to a higher risk of treatment failure and/or complications (e.g., renal transplant recipients, subjects with clinically significant persistent granulocytopenia [absolute neutrophil count <1000/microliter (µL)], and subjects receiving immunosuppressive therapy, including corticosteroid therapy [>40 mg/day prednisolone or equivalent for >1 week or >=20 milligrams per day (mg/day) prednisolone or equivalent for >6 weeks; or prednisolone or equivalent >=10 mg/day for >6 weeks]). Subjects with a known cluster of differentiation 4 (CD4) count of <200 cells/mm^3 should not be enrolled.
* The subject has uncontrolled diabetes, defined as a non-fasting glucose value >300 milligrams per deciliter (mg/dL) or based on investigator judgment.
* The subject has any of the following: A medical condition that requires medication that may be aggravated by inhibition of acetylcholinesterase, such as: a) Poorly controlled asthma or chronic obstructive pulmonary disease at Baseline and, in the opinion of the investigator, not stable on current therapy; b) Acute severe pain, uncontrolled with conventional medical management; c) Active peptic ulcer disease; d) Parkinson disease; e) Myasthenia gravis; f) A history of seizure disorder requiring medications for control (this does not include a history of childhood febrile seizures) OR Any surgical or medical condition (active or chronic) that may interfere with drug absorption, distribution, metabolism, or excretion of the study drug (e.g., ileostomy or malabsorption syndrome). Subjects who have had a gastric bypass or a cholecystectomy are excluded from the study OR Hemoglobin value <12 grams per deciliter (g/dL) or a known uncorrected iron deficiency.
* The subject, in the judgment of the investigator, would not be able or willing to comply with the protocol or complete study follow-up.
* The subject has a serious underlying disease that could be imminently life threatening, or the subject is unlikely to survive for the duration of the study period.
* The subject has acute cystitis that is known or suspected to be due to fungal, parasitic, or viral pathogens; or known or suspected to be due to Pseudomonas aeruginosa or Enterobacteriaceae (other than Escherichia coli [E. coli]) as the contributing pathogen.
* The subject has symptoms known or suspected to be caused by another disease process such as asymptomatic bacteriuria or chronic interstitial cystitis.
* The subject has an anatomical or physiological anomaly that predisposes the subject to UTIs or may be a source of persistent bacterial colonization, including calculi, obstruction or stricture of the urinary tract, primary renal disease (e.g., polycystic renal disease), or neurogenic bladder, or the subject has a history of anatomical or functional abnormalities of the urinary tract (e.g., chronic vesico-ureteral reflux, detrusor insufficiency).
* The subject has an indwelling catheter, nephrostomy, ureter stent, or other foreign material in the urinary tract.
* The subject who, in the opinion of the investigator, has an otherwise complicated UTI, an active upper UTI (e.g., pyelonephritis, urosepsis), signs and symptoms onset >=96 hours before the Screening assessment, or a temperature >=101 degree Fahrenheit, flank pain, chills, or any other manifestations suggestive of upper UTI.
* The subject has anuria, oliguria, or significant impairment of renal function (creatinine clearance <30 milliliters per minute [mL/min] or clinically significant elevated serum creatinine).
* The subject presents with vaginal discharge at Baseline (e.g., suspected sexually transmitted disease).
* The subject has congenital long QT syndrome or known prolongation of the corrected QT (QTc) interval.
* The subject has uncompensated heart failure, defined as New York Heart Association Class >=III.
* The subject has severe left ventricular hypertrophy.
* The subject has a family history of QT prolongation or sudden death.
* The subject has a recent history of vasovagal syncope or episodes of symptomatic bradycardia or bradyarrhythmia within the last 12 months.
* The subject is taking QT-prolonging drugs or drugs known to increase the risk of torsades de points (TdP) per the www.crediblemeds.org "Known Risk of TdP" category at the time of her Baseline Visit, which cannot be safely discontinued from the Baseline Visit to the TOC Visit; or the subject is taking a strong cytochrome P450 enzyme 3A4 (CYP3A4) inhibitor or a strong P-glycoprotein (P-gp) inhibitor.
* The subject has a QT interval corrected for heart rate (QTc) >450 milliseconds (msec) or a QTc >480 msec for subjects with bundle-branch block.
* The subject has a known ALT value >2 times upper limit of normal (ULN).
* The subject has a known bilirubin value >1.5 times ULN (isolated bilirubin >1.5 times ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* The subject has a current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones), including symptomatic viral hepatitis or moderate-to-severe liver insufficiency (Child Pugh class B or C).
* The subject has received treatment with other systemic antimicrobials or systemic antifungals within 1 week before study entry.
* The subject must agree not to use the medications or nondrug therapies from the Baseline Visit through the TOC Visit.
* The subject has been previously enrolled in this study or has previously been treated with gepotidacin.
* The subject has participated in a clinical trial and has received an investigational product within 30 days or 5 half-lives, whichever is longer.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 22 (Actual)
Dates: Start 2018-07-23 (Actual); Primary Completion 2019-01-07 (Actual); Study Completion 2019-01-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline (for GlaxoSmithKline; Human Genome Sciences Inc., a GSK Company; Sirtris, a GSK Company; Stiefel, a GSK Company; ViiV Healthcare)
Locations (1):
- GSK Investigational Site, La Mesa, California, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=20368

REFERENCES:
- [Background] Overcash JS, Tiffany CA, Scangarella-Oman NE, Perry CR, Tao Y, Hossain M, Barth A, Dumont EF. Phase 2a Pharmacokinetic, Safety, and Exploratory Efficacy Evaluation of Oral Gepotidacin (GSK2140944) in Female Participants with Uncomplicated Urinary Tract Infection (Acute Uncomplicated Cystitis). Antimicrob Agents Chemother. 2020 Jun 23;64(7):e00199-20. doi: 10.1128/AAC.00199-20. Print 2020 Jun 23. PMID 32284384
- [Derived] Nuzzo A, Van Horn S, Traini C, Perry CR, Dumont EF, Scangarella-Oman NE, Gardiner DF, Brown JR. Microbiome recovery in adult females with uncomplicated urinary tract infections in a randomised phase 2A trial of the novel antibiotic gepotidacin (GSK140944). BMC Microbiol. 2021 Jun 15;21(1):181. doi: 10.1186/s12866-021-02245-8. PMID 34130619
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217381&parentIdentifier=206899&attachmentIdentifier=5f4d22a5-b833-491c-830b-1a2e290982f9&fileName=gsk-206899-protocol-redact.pdf&versionIdentifier=
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217381&parentIdentifier=206899&attachmentIdentifier=75c5eebb-26e9-4eeb-a18d-37bd9f3f0722&fileName=gsk-206899-reporting-and-analysis-plan-redact.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an open-label study to evaluate the pharmacokinetic (PK) of repeat oral doses of gepotidacin in adult female participants with clinical signs and symptoms of acute cystitis.
Pre-assignment Details: A total of 22 participants were enrolled in this study. This study was conducted at a single center in the United States.
Groups:
- Gepotidacin 1500 mg: All participants received gepotidacin 1500 milligram (mg) (2*750 mg, tablets), twice daily (BID), orally on Day 1 to Day 5. The total daily dose received was 3000 mg. All doses were administered after food consumption and with water.
Period: Overall Study
Arm/Group | Gepotidacin 1500 mg
Started | 22
Completed | 20
Not Completed | 2
Not completed — Family emergency | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Groups:
- Gepotidacin 1500 mg: All participants received gepotidacin 1500 mg (2*750 mg, tablets), BID, orally on Day 1 to Day 5. The total daily dose received was 3000 mg. All doses were administered after food consumption and with water.
Arm/Group | Gepotidacin 1500 mg
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.1 (12.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 4
  White - White/Caucasian/European Heritage | 18

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-time Curve (AUC) From Zero (Pre-dose) Over the Dosing Interval (AUC[0-tau]) of Gepotidacin
Description: Blood samples were collected to evaluate the PK of gepotidacin at the indicated time points. The PK parameters were calculated by standard non-compartmental analysis. PK Parameter Population consisted of all participants who received gepotidacin 1500 mg BID through the completion of all PK collections for whom valid and evaluable plasma PK parameters were derived for gepotidacin.
Time Frame: Days 1 and 4: Pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours post-dose
Population: PK Parameter Population. All the participants in the study were analyzed (22 Participants) but only those participants with data available at the specified data points were analyzed (represented by n=X in the category titles).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours* nanogram per milliliter (h*ng/mL)
Arm/Group | Gepotidacin 1500 mg
Number analyzed (Participants) | 22
Hours* nanogram per milliliter (h*ng/mL)
  Day 1, n=20: number analyzed (Participants) | 20
  Day 1, n=20 | 20236.2 (28.6)
  Day 4, n=21: number analyzed (Participants) | 21
  Day 4, n=21 | 29313.8 (31.8)

2. Primary Outcome: Maximum Plasma Concentration (Cmax) of Gepotidacin
Description: Blood samples were collected to evaluate the PK of gepotidacin at the indicated time points. The PK parameters were calculated by standard non-compartmental analysis.
Time Frame: Days 1 and 4: Pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter (ng/mL)
Arm/Group | Gepotidacin 1500 mg
Number analyzed (Participants) | 22
Nanogram per milliliter (ng/mL)
  Day 1, n=20: number analyzed (Participants) | 20
  Day 1, n=20 | 5891 (47.3)
  Day 4, n=21: number analyzed (Participants) | 21
  Day 4, n=21 | 8437 (38.0)

3. Primary Outcome: Time of Occurrence of Cmax (Tmax) of Gepotidacin
Description: as for outcome 2
Time Frame: Days 1 and 4: Pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours post-dose
Population: as for outcome 1
Measure: Median (Full Range); unit: Hours
Arm/Group | Gepotidacin 1500 mg
Number analyzed (Participants) | 22
Hours
  Day 1, n=20: number analyzed (Participants) | 20
  Day 1, n=20 | 1.500 [0.47 to 3.07]
  Day 4, n=21: number analyzed (Participants) | 21
  Day 4, n=21 | 1.917 [0.45 to 4.12]

4. Primary Outcome: Apparent Steady State Clearance (CLss/F) of Gepotidacin
Description: Blood samples were collected to evaluate the PK of gepotidacin at the indicated time points. The PK parameters were calculated by standard non-compartmental analysis. CLss/F was calculated as Dose divided by AUC(0-tau).
Time Frame: Day 4: Pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours post-dose
Population: PK Parameter Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per hour
Arm/Group | Gepotidacin 1500 mg
Number analyzed (Participants) | 21
Liters per hour | 51.17 (31.8)

5. Primary Outcome: Accumulation Ratio (Ro) of Gepotidacin
Description: Blood samples were collected to evaluate the PK of gepotidacin at the indicated time points. The PK parameters were calculated by standard non-compartmental analysis. Accumulation ratio (Ro) was calculated as ratio of AUC(0-tau) at Day 4 to AUC(0-tau) at Day 1.
Time Frame: Days 1 and 4: Pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours post-dose
Population: PK Parameter Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Gepotidacin 1500 mg
Number analyzed (Participants) | 19
Ratio | 1.402 (20.4)

6. Primary Outcome: Plasma Pre-dose Concentration (Ctau) of Gepotidacin
Description: as for outcome 2
Time Frame: Days 1 to 5: Pre-dose
Population: PK Parameter Population. Only those participants with data available at the indicated time points were analyzed (represented by n= X in the category titles).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Gepotidacin 1500 mg
Number analyzed (Participants) | 22
ng/mL
  Day 1, Pre-dose, n=22 | NA (NA) — Data was not available as all concentration values were below the lower limit of quantification.
  Day 2, Pre-dose, n=21: number analyzed (Participants) | 21
  Day 2, Pre-dose, n=21 | 620.5 (62.3)
  Day 3, Pre-dose, n=21: number analyzed (Participants) | 21
  Day 3, Pre-dose, n=21 | 789.3 (37.4)
  Day 4, Pre-dose, n=21: number analyzed (Participants) | 21
  Day 4, Pre-dose, n=21 | 851.4 (41.4)
  Day 5, Pre-dose, n=21: number analyzed (Participants) | 21
  Day 5, Pre-dose, n=21 | 818.9 (46.4)

7. Secondary Outcome: Amount of Drug Excreted Over 12 Hours (Ae12hours) of Gepotidacin
Description: Urine samples were collected to evaluate the PK of gepotidacin at the indicated time points. The PK parameters were calculated by standard non-compartmental analysis. Ae12hours was calculated by adding all the fractions of drug collected over all the allotted time intervals.
Time Frame: Days 1 and 4: Pre-dose and at 0 to 2 hours, 2 to 4 hours, 4 to 6 hours, 6 to 8 hours, 8 to 10 hours, and 10 to 12 hours post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg
Arm/Group | Gepotidacin 1500 mg
Number analyzed (Participants) | 22
mg
  Day 1, n=20: number analyzed (Participants) | 20
  Day 1, n=20 | 298.7 (107.6)
  Day 4, n=21: number analyzed (Participants) | 21
  Day 4, n=21 | 460.0 (55.8)

8. Secondary Outcome: Amount of Drug Excreted in Urine in a Time Interval (Ae[t1-t2]) of Gepotidacin
Description: Ae(t1-t2) measure the amount of drug excreted in urine in a time intervals 0 to 2 hours, 2 to 4 hours, 4 to 6 hours, 6 to 8 hours, 8 to 10 hours, and 10 to 12 hours post-dose on Days 1 and 4. The PK parameters were calculated by standard non-compartmental analysis.
Time Frame: as for outcome 7
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg
Arm/Group | Gepotidacin 1500 mg
Number analyzed (Participants) | 22
mg
  Day 1, Ae (0-2),n=17: number analyzed (Participants) | 17
  Day 1, Ae (0-2),n=17 | NA (NA) — Data was not available as all concentration values were below the lower limit of quantification.
  Day 4, Ae (0-2),n=18: number analyzed (Participants) | 18
  Day 4, Ae (0-2),n=18 | 63.05 (151.7)
  Day 1, Ae (2-4),n=17: number analyzed (Participants) | 17
  Day 1, Ae (2-4),n=17 | 131.9 (59.5)
  Day 4, Ae (2-4),n=12: number analyzed (Participants) | 12
  Day 4, Ae (2-4),n=12 | 168.1 (96.5)
  Day 1, Ae (4-6) ,n=14: number analyzed (Participants) | 14
  Day 1, Ae (4-6) ,n=14 | 87.01 (90.0)
  Day 4, Ae (4-6),n=18: number analyzed (Participants) | 18
  Day 4, Ae (4-6),n=18 | 128.6 (96.8)
  Day 1, Ae (6-8),n=16: number analyzed (Participants) | 16
  Day 1, Ae (6-8),n=16 | 54.60 (72.1)
  Day 4, Ae (6-8),n=17: number analyzed (Participants) | 17
  Day 4, Ae (6-8),n=17 | 84.08 (92.0)
  Day 1, Ae (8-10),n=9: number analyzed (Participants) | 9
  Day 1, Ae (8-10),n=9 | 18.51 (49.9)
  Day 4, Ae (8-10),n=10: number analyzed (Participants) | 10
  Day 4, Ae (8-10),n=10 | 34.68 (69.2)
  Day 1, Ae (10-12),n=14: number analyzed (Participants) | 14
  Day 1, Ae (10-12),n=14 | 18.03 (151.2)
  Day 4, Ae (10-12),n=15: number analyzed (Participants) | 15
  Day 4, Ae (10-12),n=15 | 32.77 (83.5)

9. Secondary Outcome: Percentage of the Given Dose of Drug Excreted in Urine (fe%) of Gepotidacin
Description: Urine samples were collected to evaluate the PK of gepotidacin at the indicated time points. fe% was calculated as fe% = (Ae 12 hours/Dose) multiply by 100. The PK parameters were calculated by standard non-compartmental analysis.
Time Frame: as for outcome 7
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of dose
Arm/Group | Gepotidacin 1500 mg
Number analyzed (Participants) | 22
Percentage of dose
  Day 1, n=20: number analyzed (Participants) | 20
  Day 1, n=20 | 19.91 (107.6)
  Day 4, n=21: number analyzed (Participants) | 21
  Day 4, n=21 | 30.67 (55.8)

10. Secondary Outcome: Renal Clearance (CLr) of Gepotidacin
Description: Urine samples were collected to evaluate the PK of gepotidacin at the indicated time points. CLr was calculated as CLr = Ae 12 hours/AUC(0-tau). The PK parameters were calculated by standard non-compartmental analysis.
Time Frame: as for outcome 7
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per hour
Arm/Group | Gepotidacin 1500 mg
Number analyzed (Participants) | 22
Liters per hour
  Day 1, n=20: number analyzed (Participants) | 20
  Day 1, n=20 | 14.76 (118.2)
  Day 4, n=21: number analyzed (Participants) | 21
  Day 4, n=21 | 15.69 (45.2)

11. Secondary Outcome: Urine Pre-dose Concentration (Ctau) of Gepotidacin
Description: Urine samples were collected to evaluate the PK of gepotidacin at the indicated time points. The PK parameters were calculated by standard non-compartmental analysis.
Time Frame: Days 1 to 5: Pre-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | Gepotidacin 1500 mg
Number analyzed (Participants) | 22
Micrograms per milliliter
  Day 1, Pre-dose, n=21: number analyzed (Participants) | 21
  Day 1, Pre-dose, n=21 | NA (NA) — Data was not available as all concentration values were below the lower limit of quantification.
  Day 2, Pre-dose, n=20: number analyzed (Participants) | 20
  Day 2, Pre-dose, n=20 | 279.1 (154.7)
  Day 3, Pre-dose, n=21: number analyzed (Participants) | 21
  Day 3, Pre-dose, n=21 | 322.2 (138.8)
  Day 4, Pre-dose, n=21: number analyzed (Participants) | 21
  Day 4, Pre-dose, n=21 | 326.7 (248.7)
  Day 5, Pre-dose, n=21: number analyzed (Participants) | 21
  Day 5, Pre-dose, n=21 | 351.7 (146.5)

12. Secondary Outcome: Number of Participants With Non-serious Adverse Events (Non-SAEs) and Serious AEs (SAEs)
Description: An AEs is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. An SAE is defined as any untoward medical occurrence that, at any dose: results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent disability/incapacity; is a congenital anomaly/birth defect; and other important medical events which may require medical or surgical intervention. Safety Population consisted of all participants who received at least 1 dose of gepotidacin.
Time Frame: Up to Day 31
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Gepotidacin 1500 mg
Number analyzed (Participants) | 22
Participants
  Non-SAEs | 21
  SAEs | 1

13. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: Vital signs including SBP and DBP were measured in semi-supine position after 5 minutes of rest for the participants in a quiet setting without distractions. Baseline was defined as the latest non-missing value at Day -1 or at Day 1 pre-dose. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value. Assessment at Test-of-cure visit was conducted between any day of Days 10 to 13.
Time Frame: Baseline, Day 2, Day 3, Day 4, Day 5 and Days 10 to 13 (Test-of-cure visit)
Population: Safety Population. Only those participants with data available at the indicated time points were analyzed (represented by n= X in the category titles).
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Gepotidacin 1500 mg
Number analyzed (Participants) | 22
Millimeters of mercury
  SBP, Day 2,n=22 | -3.1 (16.13)
  SBP, Day 3,n=22 | -0.3 (15.74)
  SBP, Day 4,n=21: number analyzed (Participants) | 21
  SBP, Day 4,n=21 | -1.5 (13.10)
  SBP, Day 5,n=21: number analyzed (Participants) | 21
  SBP, Day 5,n=21 | 0.9 (15.46)
  SBP, Days 10 to 13,n=20: number analyzed (Participants) | 20
  SBP, Days 10 to 13,n=20 | 1.5 (14.21)
  DBP, Day 2,n=22 | -2.3 (9.32)
  DBP, Day 3,n=22 | -1.1 (11.64)
  DBP, Day 4,n=21: number analyzed (Participants) | 21
  DBP, Day 4,n=21 | 0.5 (9.65)
  DBP, Day 5,n=21: number analyzed (Participants) | 21
  DBP, Day 5,n=21 | 4.7 (7.23)
  DBP, Days 10 to 13,n=20: number analyzed (Participants) | 20
  DBP, Days 10 to 13,n=20 | 2.7 (8.77)

14. Secondary Outcome: Change From Baseline in Pulse Rate
Description: Vital sign including pulse rate was measured in semi-supine position after 5 minutes of rest for the participants in a quiet setting without distractions. Baseline was defined as the latest non-missing value at Day -1 or at Day 1 pre-dose. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value. Assessment at Test-of-cure visit was conducted between any day of Days 10 to 13.
Time Frame: Baseline, Day 2, Day 3, Day 4, Day 5 and Days 10 to 13 (Test-of-cure visit)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Gepotidacin 1500 mg
Number analyzed (Participants) | 22
Beats per minute
  Day 2,n=22 | 2.2 (9.07)
  Day 3,n=22 | 2.4 (10.24)
  Day 4,n=21: number analyzed (Participants) | 21
  Day 4,n=21 | 2.9 (12.60)
  Day 5,n=21: number analyzed (Participants) | 21
  Day 5,n=21 | 7.2 (9.50)
  Days 10 to 13,n=20: number analyzed (Participants) | 20
  Days 10 to 13,n=20 | 0.8 (12.38)

15. Secondary Outcome: Change From Baseline in Body Temperature
Description: Vital sign including body temperature was measured in semi-supine position after 5 minutes of rest for the participants in a quiet setting without distractions. Baseline was defined as the latest non-missing value at Day -1 or at Day 1 pre-dose. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value. Assessment at Test-of-cure visit was conducted between any day of Days 10 to 13.
Time Frame: Baseline, Day 2, Day 3, Day 4, Day 5 and Days 10 to 13 (Test-of-cure visit)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Degree Celsius
Arm/Group | Gepotidacin 1500 mg
Number analyzed (Participants) | 22
Degree Celsius
  Day 2,n=22 | -0.05 (0.246)
  Day 3,n=22 | -0.06 (0.292)
  Day 4,n=21: number analyzed (Participants) | 21
  Day 4,n=21 | 0.02 (0.405)
  Day 5,n=21: number analyzed (Participants) | 21
  Day 5,n=21 | -0.05 (0.287)
  Days 10 to 13,n=20: number analyzed (Participants) | 20
  Days 10 to 13,n=20 | -0.10 (0.270)

16. Secondary Outcome: Change From Baseline in Electrocardiogram (ECG) Parameters: PR Interval, QRS Duration, QT Interval, Corrected QT Interval Using Bazett's Formula (QTcB) and Corrected QT Interval Using Fridericia's Formula (QTcF)
Description: A 12-lead ECG was measured in semi-supine position using an ECG machine that measured PR interval, QRS duration, QT interval, QTcB and QTcF. Baseline was defined as the latest non-missing value at Day -1 or at Day 1 pre-dose. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value.
Time Frame: Baseline; Day 1: 2 hours; Day 4: pre-dose and 2 hours
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Millisecond
Arm/Group | Gepotidacin 1500 mg
Number analyzed (Participants) | 22
Millisecond
  PR interval, Day 1: 2 hours, n=22 | -1.9 (11.34)
  PR interval, Day 4: pre-dose,n=21: number analyzed (Participants) | 21
  PR interval, Day 4: pre-dose,n=21 | 0.1 (14.56)
  PR interval, Day 4: 2 hours,n=21: number analyzed (Participants) | 21
  PR interval, Day 4: 2 hours,n=21 | -3.5 (10.17)
  QRS duration, Day 1: 2 hours, n=22 | -0.7 (8.32)
  QRS duration, Day 4: pre-dose,n=21: number analyzed (Participants) | 21
  QRS duration, Day 4: pre-dose,n=21 | -0.9 (4.10)
  QRS duration, Day 4: 2 hours,n=21: number analyzed (Participants) | 21
  QRS duration, Day 4: 2 hours,n=21 | 2.1 (4.29)
  QT interval, Day 1: 2 hours, n=22 | 15.0 (21.56)
  QT interval, Day 4: pre-dose,n=21: number analyzed (Participants) | 21
  QT interval, Day 4: pre-dose,n=21 | -5.4 (26.86)
  QT interval, Day 4: 2 hours,n=21: number analyzed (Participants) | 21
  QT interval, Day 4: 2 hours,n=21 | 8.7 (27.46)
  QTcB interval, Day 1: 2 hours, n=22 | 4.5 (14.37)
  QTcB interval, Day 4: pre-dose,n=21: number analyzed (Participants) | 21
  QTcB interval, Day 4: pre-dose,n=21 | -6.2 (17.25)
  QTcB interval, Day 4: 2 hours,n=21: number analyzed (Participants) | 21
  QTcB interval, Day 4: 2 hours,n=21 | 0.4 (27.33)
  QTcF interval, Day 1: 2 hours, n=22 | 8.2 (14.45)
  QTcF interval, Day 4: pre-dose,n=21: number analyzed (Participants) | 21
  QTcF interval, Day 4: pre-dose,n=21 | -5.8 (17.57)
  QTcF interval, Day 4: 2 hours,n=21: number analyzed (Participants) | 21
  QTcF interval, Day 4: 2 hours,n=21 | 3.4 (24.84)

17. Secondary Outcome: Change From Baseline in Hematology Parameters: Basophils, Eosinophils, Lymphocytes, Monocytes, Neutrophils and Platelet Counts
Description: Blood samples were collected to analyze the hematology parameters: Basophils, Eosinophils, Lymphocytes, Monocytes, Neutrophils and Platelet counts. Baseline was defined as Day -1. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value. Assessment at Test-of-cure visit was conducted between any day of Days 10 to 13.
Time Frame: Baseline, Day 3, Day 5 and Days 10 to 13 (Test-of-cure visit)
Population: Safety Population. All the participants in the study were analyzed (22 Participants) but only those participants with data available at the specified data points were analyzed (represented by n=X in the category titles).
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | Gepotidacin 1500 mg
Number analyzed (Participants) | 22
10^9 cells per liter
  Day 3, Basophils, n=16: number analyzed (Participants) | 16
  Day 3, Basophils, n=16 | 0.013 (0.0652)
  Day 5, Basophils, n=14: number analyzed (Participants) | 14
  Day 5, Basophils, n=14 | -0.003 (0.0164)
  Days 10 to 13, Basophils, n=15: number analyzed (Participants) | 15
  Days 10 to 13, Basophils, n=15 | 0.000 (0.0146)
  Day 3, Eosinophils, n=18: number analyzed (Participants) | 18
  Day 3, Eosinophils, n=18 | 0.013 (0.0550)
  Day 5, Eosinophils, n=17: number analyzed (Participants) | 17
  Day 5, Eosinophils, n=17 | -0.003 (0.0969)
  Days 10 to 13, Eosinophils, n=16: number analyzed (Participants) | 16
  Days 10 to 13, Eosinophils, n=16 | 0.051 (0.0492)
  Day 3, Lymphocytes, n=19: number analyzed (Participants) | 19
  Day 3, Lymphocytes, n=19 | 0.039 (0.5201)
  Day 5, Lymphocytes, n=18: number analyzed (Participants) | 18
  Day 5, Lymphocytes, n=18 | 0.041 (0.4856)
  Days 10 to 13, Lymphocytes, n=17: number analyzed (Participants) | 17
  Days 10 to 13, Lymphocytes, n=17 | 0.232 (0.4001)
  Day 3, Monocytes, n=19: number analyzed (Participants) | 19
  Day 3, Monocytes, n=19 | -0.053 (0.1080)
  Day 5, Monocytes, n=18: number analyzed (Participants) | 18
  Day 5, Monocytes, n=18 | -0.069 (0.1468)
  Days 10 to 13, Monocytes, n=17: number analyzed (Participants) | 17
  Days 10 to 13, Monocytes, n=17 | -0.039 (0.1415)
  Day 3, Neutrophils, n=19: number analyzed (Participants) | 19
  Day 3, Neutrophils, n=19 | -0.673 (1.9611)
  Day 5, Neutrophils, n=18: number analyzed (Participants) | 18
  Day 5, Neutrophils, n=18 | -0.948 (2.3174)
  Days 10 to 13, Neutrophils, n=17: number analyzed (Participants) | 17
  Days 10 to 13, Neutrophils, n=17 | -0.841 (1.4779)
  Day 3, Platelet counts, n=19: number analyzed (Participants) | 19
  Day 3, Platelet counts, n=19 | -3.6 (22.94)
  Day 5, Platelet counts, n=18: number analyzed (Participants) | 18
  Day 5, Platelet counts, n=18 | 7.8 (32.33)
  Days 10 to 13, Platelet counts, n=17: number analyzed (Participants) | 17
  Days 10 to 13, Platelet counts, n=17 | 3.7 (33.59)

18. Secondary Outcome: Change From Baseline in Hematology Parameter: Hemoglobin
Description: Blood samples were collected to analyze the hematology parameter: Hemoglobin. Baseline was defined as Day -1. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value. Assessment at Test-of-cure visit was conducted between any day of Days 10 to 13.
Time Frame: Baseline, Day 3, Day 5 and Days 10 to 13 (Test-of-cure visit)
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Gepotidacin 1500 mg
Number analyzed (Participants) | 22
Grams per liter
  Day 3, n=19: number analyzed (Participants) | 19
  Day 3, n=19 | -3.4 (8.15)
  Day 5, n=18: number analyzed (Participants) | 18
  Day 5, n=18 | -0.6 (9.34)
  Days 10 to 13, n=17: number analyzed (Participants) | 17
  Days 10 to 13, n=17 | -8.2 (7.40)

19. Secondary Outcome: Change From Baseline in Hematology Parameter: Hematocrit
Description: Blood samples were collected to analyze the hematology parameter: Hematocrit. Baseline was defined as Day -1. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value. Assessment at Test-of-cure visit was conducted between any day of Days 10 to 13.
Time Frame: Baseline, Day 3, Day 5 and Days 10 to 13 (Test-of-cure visit)
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Percentage of red blood cells in blood
Arm/Group | Gepotidacin 1500 mg
Number analyzed (Participants) | 22
Percentage of red blood cells in blood
  Day 3, n=19: number analyzed (Participants) | 19
  Day 3, n=19 | 0.75 (3.186)
  Day 5, n=18: number analyzed (Participants) | 18
  Day 5, n=18 | -0.54 (3.643)
  Days 10 to 13, n=17: number analyzed (Participants) | 17
  Days 10 to 13, n=17 | -2.30 (2.956)

20. Secondary Outcome: Change From Baseline in Hematology Parameter: Erythrocyte Mean Corpuscular Hemoglobin
Description: Blood samples were collected to analyze the hematology parameter: Erythrocyte Mean Corpuscular Hemoglobin. Baseline was defined as Day -1. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value. Assessment at Test-of-cure visit was conducted between any day of Days 10 to 13.
Time Frame: Baseline, Day 3, Day 5 and Days 10 to 13 (Test-of-cure visit)
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Picogram
Arm/Group | Gepotidacin 1500 mg
Number analyzed (Participants) | 22
Picogram
  Day 3, n=19: number analyzed (Participants) | 19
  Day 3, n=19 | 0.13 (0.564)
  Day 5, n=18: number analyzed (Participants) | 18
  Day 5, n=18 | 0.03 (0.465)
  Days 10 to 13, n=17: number analyzed (Participants) | 17
  Days 10 to 13, n=17 | 0.16 (0.348)

21. Secondary Outcome: Change From Baseline in Hematology Parameter: Erythrocyte Mean Corpuscular Volume
Description: Blood samples were collected to analyze the hematology parameter: Erythrocyte Mean Corpuscular Volume. Baseline was defined as Day -1. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value. Assessment at Test-of-cure visit was conducted between any day of Days 10 to 13.
Time Frame: Baseline, Day 3, Day 5 and Days 10 to 13 (Test-of-cure visit)
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Femtoliter
Arm/Group | Gepotidacin 1500 mg
Number analyzed (Participants) | 22
Femtoliter
  Day 3, n=19: number analyzed (Participants) | 19
  Day 3, n=19 | 4.53 (5.814)
  Day 5, n=18: number analyzed (Participants) | 18
  Day 5, n=18 | -0.72 (4.668)
  Days 10 to 13, n=17: number analyzed (Participants) | 17
  Days 10 to 13, n=17 | 1.14 (6.252)

22. Secondary Outcome: Change From Baseline in Hematology Parameter: Red Blood Cell Count
Description: Blood samples were collected to analyze the hematology parameter: Red blood cell count. Baseline was defined as Day -1. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value. Assessment at Test-of-cure visit was conducted between any day of Days 10 to 13.
Time Frame: Baseline, Day 3, Day 5 and Days 10 to 13 (Test-of-cure visit)
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter
Arm/Group | Gepotidacin 1500 mg
Number analyzed (Participants) | 22
10^12 cells per liter
  Day 3, n=19: number analyzed (Participants) | 19
  Day 3, n=19 | -0.135 (0.2574)
  Day 5, n=18: number analyzed (Participants) | 18
  Day 5, n=18 | -0.031 (0.3060)
  Days 10 to 13, n=17: number analyzed (Participants) | 17
  Days 10 to 13, n=17 | -0.298 (0.2552)

23. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters: Albumin and Protein
Description: Blood samples were collected to analyze the chemistry parameters: Albumin and Protein. Baseline was defined as Day -1. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value. Assessment at Test-of-cure visit was conducted between any day of Days 10 to 13.
Time Frame: Baseline, Day 3, Day 5 and Days 10 to 13 (Test-of-cure visit)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Gepotidacin 1500 mg
Number analyzed (Participants) | 22
Grams per liter
  Albumin: Day 3, n=22 | -2.0 (2.45)
  Albumin: Day 5, n=21: number analyzed (Participants) | 21
  Albumin: Day 5, n=21 | -1.4 (2.71)
  Albumin: Days 10 to 13, n=20: number analyzed (Participants) | 20
  Albumin: Days 10 to 13, n=20 | -1.3 (2.90)
  Protein: Day 3, n=22 | -3.0 (3.82)
  Protein: Day 5, n=21: number analyzed (Participants) | 21
  Protein: Day 5, n=21 | -2.6 (4.52)
  Protein: Days 10 to 13, n=20: number analyzed (Participants) | 20
  Protein: Days 10 to 13, n=20 | -2.4 (5.13)

24. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters: Creatinine and Bilirubin
Description: Blood samples were collected to analyze the chemistry parameters: Creatinine and Bilirubin. Baseline was defined as Day -1. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value. Assessment at Test-of-cure visit was conducted between any day of Days 10 to 13.
Time Frame: Baseline, Day 3, Day 5 and Days 10 to 13 (Test-of-cure visit)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Gepotidacin 1500 mg
Number analyzed (Participants) | 22
Micromoles per liter
  Creatinine: Day 3, n=22 | 2.411 (9.9048)
  Creatinine: Day 5, n=21: number analyzed (Participants) | 21
  Creatinine: Day 5, n=21 | 1.684 (7.7162)
  Creatinine: Days 10 to 13, n=20: number analyzed (Participants) | 20
  Creatinine: Days 10 to 13, n=20 | 0.442 (7.2981)
  Bilirubin: Day 3, n=14: number analyzed (Participants) | 14
  Bilirubin: Day 3, n=14 | -1.8932 (4.06405)
  Bilirubin: Day 5, n=15: number analyzed (Participants) | 15
  Bilirubin: Day 5, n=15 | -1.6986 (3.41356)
  Bilirubin: Days 10 to 13, n=14: number analyzed (Participants) | 14
  Bilirubin: Days 10 to 13, n=14 | -1.6856 (3.42845)

25. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters: Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST) and Alkaline Phosphatase (ALP)
Description: Blood samples were collected to analyze the chemistry parameters: ALT, AST and ALP. Baseline was defined as Day -1. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value. Assessment at Test-of-cure visit was conducted between any day of Days 10 to 13.
Time Frame: Baseline, Day 3, Day 5 and Days 10 to 13 (Test-of-cure visit)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: International units per liter
Arm/Group | Gepotidacin 1500 mg
Number analyzed (Participants) | 22
International units per liter
  ALT: Day 3, n=22 | -1.5 (4.99)
  ALT: Day 5, n=21: number analyzed (Participants) | 21
  ALT: Day 5, n=21 | 1.7 (7.51)
  ALT: Days 10 to 13, n=20: number analyzed (Participants) | 20
  ALT: Days 10 to 13, n=20 | 1.7 (7.44)
  AST: Day 3, n=22 | -1.3 (3.22)
  AST: Day 5, n=21: number analyzed (Participants) | 21
  AST: Day 5, n=21 | 1.3 (3.77)
  AST: Days 10 to 13, n=20: number analyzed (Participants) | 20
  AST: Days 10 to 13, n=20 | 2.1 (3.22)
  ALP: Day 3, n=22 | -3.3 (7.91)
  ALP: Day 5, n=21: number analyzed (Participants) | 21
  ALP: Day 5, n=21 | -4.3 (8.84)
  ALP: Days 10 to 13, n=20: number analyzed (Participants) | 20
  ALP: Days 10 to 13, n=20 | -4.5 (7.76)

26. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters: Glucose, Calcium, Chloride, Potassium, Sodium and Urea
Description: Blood samples were collected to analyze the chemistry parameters: Glucose, Calcium, Chloride, Potassium, Sodium and Urea. Baseline was defined as Day -1. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value. Assessment at Test-of-cure visit was conducted between any day of Days 10 to 13.
Time Frame: Baseline, Day 3, Day 5 and Days 10 to 13 (Test-of-cure visit)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Gepotidacin 1500 mg
Number analyzed (Participants) | 22
Millimoles per liter
  Day 3, Glucose, n=22 | 0.13121 (1.237031)
  Day 5, Glucose, n=21: number analyzed (Participants) | 21
  Day 5, Glucose, n=21 | 0.87495 (1.382514)
  Days 10 to 13, Glucose, n=20: number analyzed (Participants) | 20
  Days 10 to 13, Glucose, n=20 | -0.05274 (0.498607)
  Day 3, Calcium, n=22 | -0.05330 (0.075175)
  Day 5, Calcium, n=21: number analyzed (Participants) | 21
  Day 5, Calcium, n=21 | -0.05228 (0.093648)
  Days 10 to 13, Calcium, n=20: number analyzed (Participants) | 20
  Days 10 to 13, Calcium, n=20 | -0.07110 (0.095536)
  Day 3, Chloride, n=22 | 0.5 (2.42)
  Day 5, Chloride, n=21: number analyzed (Participants) | 21
  Day 5, Chloride, n=21 | 0.3 (2.90)
  Days 10 to 13, Chloride, n=20: number analyzed (Participants) | 20
  Days 10 to 13, Chloride, n=20 | 0.3 (2.15)
  Day 3, Potassium, n=22 | 0.04 (0.359)
  Day 5, Potassium, n=21: number analyzed (Participants) | 21
  Day 5, Potassium, n=21 | -0.05 (0.425)
  Days 10 to 13, Potassium, n=20: number analyzed (Participants) | 20
  Days 10 to 13, Potassium, n=20 | 0.01 (0.419)
  Day 3, Sodium, n=22 | -0.7 (2.29)
  Day 5, Sodium, n=21: number analyzed (Participants) | 21
  Day 5, Sodium, n=21 | -1.6 (2.13)
  Days 10 to 13, Sodium, n=20: number analyzed (Participants) | 20
  Days 10 to 13, Sodium, n=20 | -0.9 (1.65)
  Day 3, Urea, n=22 | 0.1298 (1.15836)
  Day 5, Urea, n=21: number analyzed (Participants) | 21
  Day 5, Urea, n=21 | 0.0680 (1.06275)
  Days 10 to 13, Urea, n=20: number analyzed (Participants) | 20
  Days 10 to 13, Urea, n=20 | 0.3927 (1.18063)

27. Secondary Outcome: Number of Participants With Urinalysis Dipstick Results: Glucose and Nitrites
Description: Urine samples were collected at indicated time points to analyze parameters including glucose and nitrites by dipstick. The dipstick test gives results in a semi-quantitative manner, and results for urinalysis parameters can be read as negative and positive in the urine sample. Baseline was defined as Day -1. Assessment at Test-of-cure visit was conducted between any day of Days 10 to 13. Only categories with significant values have been presented.
Time Frame: Baseline, Day 3, Day 5 and Days 10 to 13 (Test-of-cure visit)
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Gepotidacin 1500 mg
Number analyzed (Participants) | 22
Participants
  Baseline:Glucose,Negative,n=22 | 22
  Day 3:Glucose,Negative,n=22 | 22
  Day 5:Glucose,Negative,n=21: number analyzed (Participants) | 21
  Day 5:Glucose,Negative,n=21 | 21
  Days 10 to 13:Glucose,Negative,n=20: number analyzed (Participants) | 20
  Days 10 to 13:Glucose,Negative,n=20 | 20
  Baseline: Nitrites,Negative,n=22 | 13
  Baseline: Nitrites,Positive,n=22 | 9
  Day 3: Nitrites,Negative,n=22 | 22
  Day 5: Nitrites,Negative,n=21: number analyzed (Participants) | 21
  Day 5: Nitrites,Negative,n=21 | 21
  Days 10 to 13: Nitrites,Negative,n=20: number analyzed (Participants) | 20
  Days 10 to 13: Nitrites,Negative,n=20 | 20

28. Secondary Outcome: Number of Participants With Urinalysis Dipstick Results: Ketones
Description: Urine samples were collected at indicated time points to analyze parameter including ketones by dipstick. The dipstick test gives results in a semi-quantitative manner, and results for urinalysis parameters can be read as negative, 5 indicates 5 milligrams per deciliter (mg/dL) and 20 indicates 20 mg/dL in the urine sample. Baseline was defined as Day -1. Assessment at Test-of-cure visit was conducted between any day of Days 10 to 13. Only categories with significant values have been presented.
Time Frame: Baseline, Day 3, Day 5 and Days 10 to 13 (Test-of-cure visit)
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Gepotidacin 1500 mg
Number analyzed (Participants) | 22
Participants
  Baseline:Ketones,Negative,n=22 | 21
  Baseline:Ketones,20,n=22 | 1
  Day 3:Ketones,Negative,n=22 | 22
  Day 5:Ketones,Negative,n=21: number analyzed (Participants) | 21
  Day 5:Ketones,Negative,n=21 | 21
  Days 10 to 13:Ketones,Negative,n=20: number analyzed (Participants) | 20
  Days 10 to 13:Ketones,Negative,n=20 | 18
  Days 10 to 13:Ketones,5,n=20: number analyzed (Participants) | 20
  Days 10 to 13:Ketones,5,n=20 | 2

29. Secondary Outcome: Number of Participants With Urinalysis Dipstick Results: Leukocyte Esterase
Description: Urine samples were collected at indicated time points to analyze parameter including leukocyte esterase by dipstick. The dipstick test gives results in a semi-quantitative manner, and results for urinalysis parameters can be read as negative, Trace indicates 15 Leukocytes per microliter (Leuko/mcL), Small indicates 70 Leuko/mcL, Moderate indicates 125 Leuko/mcL and Large indicates 500 Leuko/mcL in the urine sample. Baseline was defined as Day -1. Assessment at Test-of-cure visit was conducted between any day of Days 10 to 13. Only categories with significant values have been presented.
Time Frame: Baseline, Day 3, Day 5 and Days 10 to 13 (Test-of-cure visit)
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Gepotidacin 1500 mg
Number analyzed (Participants) | 22
Participants
  Baseline:Leukocyte esterase,Negative,n=22 | 4
  Baseline:Leukocyte esterase,Trace,n=22 | 2
  Baseline:Leukocyte esterase,Small,n=22 | 4
  Baseline:Leukocyte esterase,Moderate,n=22 | 1
  Baseline:Leukocyte esterase,Large,n=22 | 11
  Day 3:Leukocyte esterase,Negative,n=22 | 19
  Day 3:Leukocyte esterase,Small,n=22 | 1
  Day 3:Leukocyte esterase,Moderate,n=22 | 2
  Day 5:Leukocyte esterase,Negative,n=21: number analyzed (Participants) | 21
  Day 5:Leukocyte esterase,Negative,n=21 | 16
  Day 5:Leukocyte esterase,Trace,n=21: number analyzed (Participants) | 21
  Day 5:Leukocyte esterase,Trace,n=21 | 4
  Day 5:Leukocyte esterase,Small,n=21: number analyzed (Participants) | 21
  Day 5:Leukocyte esterase,Small,n=21 | 1
  Days 10 to 13:Leukocyte esterase,Negative,n=20: number analyzed (Participants) | 20
  Days 10 to 13:Leukocyte esterase,Negative,n=20 | 19
  Days 10 to 13:Leukocyte esterase,Trace,n=20: number analyzed (Participants) | 20
  Days 10 to 13:Leukocyte esterase,Trace,n=20 | 1

30. Secondary Outcome: Number of Participants With Urinalysis Dipstick Results: Occult Blood
Description: Urine samples were collected at indicated time points to analyze parameter including occult blood by dipstick. The dipstick test gives results in a semi-quantitative manner, and results for urinalysis parameters can be read as negative, Small indicates 25 Erythrocytes per microliter (Ery/mcL), Moderate indicates 50 Ery/mcL and Large indicates 250 Ery/mcL in the urine sample. Baseline was defined as Day -1. Assessment at Test-of-cure visit was conducted between any day of Days 10 to 13. Only categories with significant values have been presented.
Time Frame: Baseline, Day 3, Day 5 and Days 10 to 13 (Test-of-cure visit)
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Gepotidacin 1500 mg
Number analyzed (Participants) | 22
Participants
  Baseline:Occult blood,Negative,n=22 | 6
  Baseline:Occult blood,Small,n=22 | 10
  Baseline:Occult blood,Moderate,n=22 | 3
  Baseline:Occult blood,Large,n=22 | 3
  Day 3:Occult blood,Negative,n=22 | 19
  Day 3:Occult blood,Small,n=22 | 1
  Day 3:Occult blood,Moderate,n=22 | 1
  Day 3:Occult blood,Large,n=22 | 1
  Day 5:Occult blood,Negative,n=21: number analyzed (Participants) | 21
  Day 5:Occult blood,Negative,n=21 | 17
  Day 5:Occult blood,Small,n=21: number analyzed (Participants) | 21
  Day 5:Occult blood,Small,n=21 | 2
  Day 5:Occult blood,Moderate,n=21: number analyzed (Participants) | 21
  Day 5:Occult blood,Moderate,n=21 | 2
  Days 10 to 13:Occult blood,Negative,n=20: number analyzed (Participants) | 20
  Days 10 to 13:Occult blood,Negative,n=20 | 18
  Days 10 to 13:Occult blood,Small,n=20: number analyzed (Participants) | 20
  Days 10 to 13:Occult blood,Small,n=20 | 2

31. Secondary Outcome: Number of Participants With Urinalysis Dipstick Results: Protein
Description: Urine samples were collected at indicated time points to analyze parameter including protein by dipstick. The dipstick test gives results in a semi-quantitative manner, and results for urinalysis parameters can be read as negative indicates <10 mg/dL, 1+ indicates 30 mg/dL and 2+ indicates 100 mg/dL in the urine sample. Baseline was defined as Day -1. Assessment at Test-of-cure visit was conducted between any day of Days 10 to 13. Only categories with significant values have been presented.
Time Frame: Baseline, Day 3, Day 5 and Days 10 to 13 (Test-of-cure visit)
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Gepotidacin 1500 mg
Number analyzed (Participants) | 22
Participants
  Baseline: Protein,Negative,n=22 | 11
  Baseline: Protein,1+,n=22 | 10
  Baseline: Protein,2+,n=22 | 1
  Day 3: Protein,Negative,n=22 | 18
  Day 3: Protein,1+,n=22 | 4
  Day 5: Protein,Negative,n=21: number analyzed (Participants) | 21
  Day 5: Protein,Negative,n=21 | 16
  Day 5: Protein,1+,n=21: number analyzed (Participants) | 21
  Day 5: Protein,1+,n=21 | 5
  Days 10 to 13: Protein,Negative,n=20: number analyzed (Participants) | 20
  Days 10 to 13: Protein,Negative,n=20 | 18
  Days 10 to 13: Protein,1+,n=20: number analyzed (Participants) | 20
  Days 10 to 13: Protein,1+,n=20 | 2

32. Secondary Outcome: Number of Participants With Abnormal Physical Examination Findings
Description: Physical examinations included assessments of the respiratory, cardiovascular, abdominal, gastrointestinal, neurological and urogenital systems. This analysis was planned but data was not collected and captured in the database.
Time Frame: Up to Day 31
Population: Safety Population. This analysis was planned but data was not collected and captured in the database.
Arm/Group | Gepotidacin 1500 mg
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Non-SAEs and SAEs were collected from start of the treatment (Day 1) up to Day 31
Description: Safety Population consisted of all participants who received at least 1 dose of gepotidacin.
Arm/Group | Gepotidacin 1500 mg
All-Cause Mortality (participants affected / at risk) | 0/22
Serious Adverse Events (participants affected / at risk) | 1/22
Other Adverse Events (participants affected / at risk) | 21/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gepotidacin 1500 mg (N=22)
Major depression (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gepotidacin 1500 mg (N=22)
Diarrhoea (Gastrointestinal disorders) | 18 (22)
Nausea (Gastrointestinal disorders) | 17 (18)
Vomiting (Gastrointestinal disorders) | 5 (5)
Viral upper respiratory tract infection (Infections and infestations) | 2 (2)
Vulvovaginal mycotic infection (Infections and infestations) | 2 (2)
Headache (Nervous system disorders) | 5 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Chest discomfort (General disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-05-10): https://cdn.clinicaltrials.gov/large-docs/42/NCT03568942/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-14): https://cdn.clinicaltrials.gov/large-docs/42/NCT03568942/SAP_001.pdf